CLINICAL TRIAL: NCT03338257
Title: Husky Reads Evaluation: Measuring Changes in Fruit and Vegetable Recognition and Liking
Brief Title: Husky Reads Effectiveness in Increasing Produce Preference and Food Group Identification in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-069-3; 601305 (Other Grant/Funding Number: CT Department of Social Services/USDA)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Childhood Obesity
Keywords: Pre-school children; fruit and vegetable acceptance; service-learning; pre-school nutrition education; childhood obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: The evaluation follows a pre-test/post-test control group design with children nested within classrooms at center and school-based early care programs located in low-income communities or areas with high SNAP eligibility rates
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Husky Reads Intervention (Experimental): The Husky Reads curriculum includes a series of 10 lessons designed to introduce preschool-age children to MyPlate while improving fruit and vegetable literacy. Each lesson includes reading at least one children's book, an activity or game, and sometimes food tasting to complement the learning objectives. Undergraduate students enrolled in the Husky Reads service-learning course at UCONN or college students participating in a paid summer internship deliver the program. Each team of 2-3 students is assigned 2-3 early care classrooms to visit and deliver Husky Reads on a weekly basis.
  Interventions: Behavioral: Husky Reads Intervention
- Wait list Control (No Intervention): Programs on the wait list for Husky Reads, participate in the pre and post intervention testing but do not receive the program.

INTERVENTIONS:
Behavioral: Husky Reads Intervention — The Husky Reads curriculum now includes a series of 10 lessons designed to introduce preschool-age children to MyPlate while improving fruit and vegetable literacy. Each lesson includes reading at least one children's book, an activity or game, and food tasting to complement learning objectives related to MyPlate and fruit/vegetable literacy. Undergraduate students enrolled in the Husky Reads service- learning course at UConn or college students participating in the paid summer internship program deliver the preschool lessons. Each team of 2-3 undergraduate students is assigned 2-3 early care classrooms to visit and deliver Husky Reads lessons to on a weekly basis.
  Arms: Husky Reads Intervention

SUMMARY:
Since 1998, UCONN undergraduate students have volunteered as part of a service- learning course to deliver a program called Husky Reads. Inspired by the nationally accepted American Academy of Pediatrics' program "Reach Out and Read," Husky Reads was first designed for promotion of health, nutrition habits and literacy by reading health-oriented books to young children in pediatric and health clinics. The Husky Reads curriculum now includes a series of 10 lessons designed to introduce preschool-age children to MyPlate while improving fruit and vegetable literacy. Undergraduate students enrolled in the Husky Reads service- learning course at UConn or college students participating in the paid summer internship program deliver the preschool lessons. Each team of 2-3 undergraduate students is assigned 2-3 early care classrooms to visit and deliver Husky Reads lessons to on a weekly basis. This series targets children at an early age because early childhood is a pivotal time to influence the path towards healthy behaviors and away from obesity. The effectiveness of the Husky Reads curriculum on a preschool age child's correct identification and liking of fruits and vegetables has not been established. The proposed evaluation uses a pre-test/post- test control group design with paired data at the child level to explore whether children who participate in Husky Reads have increased odds of correctly identifying the United States Department of Agriculture (USDA) "MyPlate" program (MyPlate) and food group concepts and trying or liking select fruits and vegetables.

DETAILED DESCRIPTION:
Since 1998, University of Connecticut (UCONN) undergraduate students have volunteered as part of a service- learning course to deliver a program called Husky Reads. Inspired by the nationally accepted American Academy of Pediatrics' program "Reach Out and Read," Husky Reads was first designed for promotion of health, nutrition habits and literacy by reading health-oriented books to young children in pediatric and health clinics. The Husky Reads curriculum now includes a series of 10 lessons designed to introduce preschool-age children to MyPlate while improving fruit and vegetable literacy. Each lesson includes reading at least one children's book, an activity or game, and food tasting to complement learning objectives related to MyPlate and fruit/vegetable literacy. Undergraduate students enrolled in the Husky Reads service- learning course at UConn or college students participating in the paid summer internship program deliver the preschool lessons. Each team of 2-3 undergraduate students is assigned 2-3 early care classrooms to visit and deliver Husky Reads lessons to on a weekly basis. This series targets children at an early age because early childhood is a pivotal time to influence the path towards healthy behaviors and away from obesity. Providing food tastings and increasing exposure to foods like fruits and vegetables is especially relevant because food preferences are developed in early childhood. Early childhood is also an important time for introducing healthy behaviors because once obesity is established in childhood; it often tracks through to adulthood and is difficult to reverse through interventions.

The effectiveness of the Husky Reads curriculum on a preschool age child's MyPlate knowledge and correct identification and liking of fruits and vegetables has not been established. A more comprehensive evaluation is needed to establish if the program is effective and contributes to quality improvement efforts. Findings from a prior evaluation suggest the ability of preschoolers to identify blueberries, strawberries, carrots and broccoli increased significantly after participation in one Husky Reads lesson. Although the findings were promising, the evaluation design lacked a control group and relied on a classroom wide assessment with hands raised as a response rather than measuring whether the ability to identify the produce items changed for a given child after participation in Husky Reads. Therefore, a more thorough evaluation of whether Husky Reads helps children learn to identify select fruits and vegetables is still needed. Questions also remain whether Husky Reads increases the odds of a child tasting and/or liking select fruits and vegetables as well as recognition of MyPlate and foods in different food groups. The proposed evaluation uses a pre-test/post- test control group design with paired data at the child level to explore whether children who participate in Husky Reads have increased odds of identifying MyPlate and food group concepts , and correctly identifying,trying or liking select fruits and vegetables.

ELIGIBILITY:
Inclusion Criteria:

* child attending center or school based early care with high family enrollment in Supplemental Nutrition Assistance (SNAP)

Exclusion Criteria:

* child whose parent has signed the "opt out" portion of the notification form.

Ages: 35 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Identification of MyPlate | Three week post 10-week intervention
  Ability to name MyPlate (Larsen et al)
Ability to place foods in MyPlate food groups | Three week post 10-week intervention
  Measured by using the Food Group Game, informed by Building a Healthy Me! evaluation survey. (Larsen et al.)
Identification of specified fruits and vegetables | Three week post 10-week intervention
  Identification using modified Carraway-Stage protocol
Preference for specified fruits and vegetables | Three week post 10-week intervention
  Fruit and vegetable liking as measured by modified Carraway-Stage protocol

CONTACTS AND LOCATIONS:
Overall Officials: Ann m Ferris, PhD, Principal Investigator — UConn Health; Erin Havens, MPH, Study Director — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
This group will share raw data with developer of testing instrument.

REFERENCES:
- [Background] Carraway-Stage V, Spangler H, Borges M, Goodell LS. Evaluation of a pictorial method to assess liking of familiar fruits and vegetables among preschool children. Appetite. 2014 Apr;75:11-20. doi: 10.1016/j.appet.2013.12.011. Epub 2013 Dec 21. PMID 24365199
- [Background] Larsen AL, Liao Y, Alberts J, Huh J, Robertson T, Dunton GF. RE-AIM Analysis of a School-Based Nutrition Education Intervention in Kindergarteners. J Sch Health. 2017 Jan;87(1):36-46. doi: 10.1111/josh.12466. PMID 27917488